CLINICAL TRIAL: NCT06987968
Title: A Phase 2, Randomized, Controlled, Open-Label, Adaptive Dose Design, Proof-of-Concept Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Two Different Dwell Times of VS-01 on Top of Standard of Care Versus Standard of Care Alone in Patients With Overt Hepatic Encephalopathy
Brief Title: A Study to See if an Investigational Medicine Called VS-01 Can Help and How Safe it is in the Treatment of Patients With Overt Hepatic Encephalopathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Genfit (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VS01_P2_24_2; 2025-521029-34-00 (Other: Other Identifier assigned by the European Medecines Agency Clinical Trials Database.)
Record Dates: First submitted 2025-05-07; First posted 2025-05-23 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Hepatic Encephalopathy; Acute on Chronic Liver Failure (ACLF); Decompensated Cirrhosis
Keywords: Liver; ammonia; toxic substances; chronic liver disease; cirrhosis; VS-01; Brain; Injury; Overt hepatic encephalopathy (OHE); Acute Decompensation (AD); Standard of Care (SOC); Acute-on-Liver Failure (ACLF)
MeSH Terms: conditions — Hepatic Encephalopathy; Acute-On-Chronic Liver Failure; Fibrosis; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VS-01 with 3 hours Dwell time+ Standard of Care (SOC) (Experimental): Patients randomized to Active Treatment group will receive VS-01 3 hours Dwell time on top of SOC
  Interventions: Drug: VS-01 on top of SOC (Active Treatment Group)
- VS-01 with 4 hours Dwell time+SOC (Experimental): Patients randomized to Active Treatment group will receive VS-01 4 hours Dwell time on top of SOC
  Interventions: Drug: VS-01 on top of SOC (Active Treatment Group)
- SOC (Other): Patients randomized to Control group will receive SOC alone
  Interventions: Drug: SOC

INTERVENTIONS:
Drug: VS-01 on top of SOC (Active Treatment Group) — Patients will received VS-01 intraperitoneally up to four consecutive days on top of SOC
  Arms: VS-01 with 3 hours Dwell time+ Standard of Care (SOC); VS-01 with 4 hours Dwell time+SOC
Drug: SOC — Patients will received SOC
  Arms: SOC

SUMMARY:
A Phase 2, Randomized, Controlled, Open-Label, Adaptive Dose Design, Proof-of-Concept Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Two Different Dwell Times of VS-01 on Top of Standard of Care versus Standard of Care Alone in Patients with Overt Hepatic Encephalopathy

ELIGIBILITY:
Inclusion Criteria:

* 1)Patients with liver cirrhosis of any underlying etiology (liver cirrhosis diagnosed by standard clinical criteria, imaging findings and/or histology), who are diagnosed with Overt hepatic encephalopathy (OHE) (according to Hepatic Encephalopathy Grading Instrument) in the presence of:

  1. Acute decompensation (AD)(defined as the onset or worsening of ascites, hepatic encephalopathy, gastrointestinal (GI) bleeding or any combination of them with or without infection); or
  2. Acute on chronic liver failure (ACLF) grade 1 according to European Association for the Study of the Liver(EASL-CLIF) criteria; 2)Presence of ascites requiring diagnostic or therapeutic paracentesis; 3)Fasting blood ammonia > upper limit of normal (ULN) at baseline (BL); 4)Patients with a dry body weight ≥40 kg and <140 kg; 5)Male and female patients ≥18 to <80 years of age on the day of signing the informed consent form (ICF); 6)Patients willing and able to provide written informed consent. If the patient is unable to fully understand or sign the written informed consent based on the Investigator's judgment, the ICF must be signed by a legal representative of the patient according to local regulation.

Exclusion Criteria:

1. ACLF grade 2 or higher as defined by European Association for the Study of the Liver-Chronic Liver Failure-Chronic Liver Failure (EASL-CLIF) criteria;
2. Presence of spontaneous or secondary bacterial peritonitis (i.e., neutrophil counts >250/mm3 in ascitic fluid);
3. Contraindication for paracentesis according to the European Association for the Study of the Liver (EASL) Clinical Practice Guidelines 2018, and American Association for the Study of Liver Diseases (AASLD)Guideline on the Treatment of Ascites, Spontaneous Bacterial Peritonitis, and Hepatorenal Syndrome 2021;
4. Alfapump® in place to manage ascites;
5. Known hypersensitivity to liposomes, history of mastocytosis, multiple hypersensitivities or similar diseases known to be associated with an increased risk of allergic/anaphylactoid reactions;
6. Upper GI bleeding within the last 7 days prior to BL, acute bleeding or bleeding upon paracentesis at Screening (SCR) or Baseline (BL);
7. Poorly controlled seizure disorder;
8. Respiratory failure requiring invasive mechanical ventilation;
9. Severe circulatory failure requiring the use of high dose vasopressors (e.g., dopamine >15 μg/kg/min, or epinephrine >0.1 μg/kg/min, or norepinephrine >0.1 μg/kg/min); the use of terlipressin or low-dose norepinephrine to treat hepatorenal syndrome is not an exclusion criterion;
10. Uncontrolled severe infection with hemodynamic instability or shock; patients may be enrolled provided anti-infectives have been administered for at least 48 hours prior to BL with an appropriate response as assessed by the Principal Investigator (PI);
11. Need for Renal replacement therapy (RRT) or any extracorporeal liver support device;
12. Any significant disease considered to be potentially detrimental or would preclude the patient from participating in and completing the study as assessed by the PI. This includes but is not limited to hepatocellular carcinoma outside Milan criteria, cholangiocarcinoma, extrahepatic cancer over the past 2 years, or people who inject drugs;
13. Individuals for whom the PI deems that study participation would be unsafe or not in the interest of the patient;
14. Pregnancy or lactation;
15. Women of childbearing potential and non-sterile male patients who are not willing to use adequate contraception from SCR to 30 days after the final dose of investigational medicinal product (IMP);
16. Participation in another interventional clinical trial within 30 days of SCR.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2025-08-25 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Time to improvement of OHE as assessed by HEGI | from randomization and up to Day 5 morning

SECONDARY OUTCOMES:
The incidence and severity ([NCI CTCAE] v5.0 grade) of treatment-emergent adverse events (TEAEs) including serious adverse events (SAEs), comprising the evaluation of vital signs, ECG parameters, and laboratory parameters | from randomization and up to Day 14 (more or less 3 days)
  [NCI CTCAE] v5.0 grade: National Cancer Institute Common Terminology Criteria for Adverse Events
Pharmacokinetics (PD) (for all arms): change from Baseline (BL) in fasting blood and peritoneal fluid ammonia levels. | from randomization up to Day 14 (more or less 3 days)
Pharmacokinetics (PK) (for active treatment arms): blood and peritoneal fluid concentration-time profile of baseline (BL) corrected citric acid and lipids in patients treated with VS-01. | From randomization up to Day 5 or EOT (only for patients treated during 4 days)

CONTACTS AND LOCATIONS:
Overall Officials: Pejvack MOTLAGH, M.D, M.Sc, Study Director — Genfit
Locations (6):
- 96 Jonathan Lucas St, CSB (Main Hospital), Suite 908, Charleston, South Carolina, United States
- Nouvel Hôpital Civil, Service de Medecine Intensive Reanimation, 1, place de l'Hôpital, Strasbourg, France
- Georgia (4):
  - Georgian Clinics" Kutaisi Referral Hospital 2, Otskheli str., Kutaisi
  - LEPL The First University Clinic of Tbilisi State, Medical University, Gudamakari str.4,,LEPL The First University Clinic, Tbilisi
  - LLC Geo Hospitals Tbilisi, Multiprofile Medical Center, Tsinandali ,str. 9/3, Tbilisi
  - Tbilisi State Medical University and Ingorokva, High Medical Technology University Clinic, Tsinandali Street, Tbilisi